CLINICAL TRIAL: NCT05351619
Title: The Effect of Implementing Oral Care Bundle on Critical Care Nurses' Practice and Mechanically Ventilated Patients' Outcomes
Brief Title: Implementing Oral Care Bundle on Critical Care Nurses' Practice and Mechanically Ventilated Patients' Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0222
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Ventilator Associated Pneumonia
Keywords: oral care bundle, Critical Care Nurses' Practice, Mechanically Ventilated Patients
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: This study will be conducted in three phases; preparation, implementation, and evaluation.
  Implementation phase
  * For nurses:
    * Nurses' demographic characteristics will be collected by using part I of tool I.
    * Critical care nurses' practice of the oral care bundle will be observed by using part II of tool I.
  * For patients:
    * An initial assessment will be carried out for all MV patients in selected ICUs on admission to confirm that they are free from exclusion criteria.
    * Patients' characteristics and health-relevant data will be collected by the PI on the first day of admission using part I of tool II.
    * Assessment of the occurrence of VAP will be done for both groups on the first, third, and sixth days of the patient's admission to the ICU by using part II of tool II.
    * An oral assessment scale will be carried out for both groups on the first, third, and sixth days of patient admission by using part III of tool II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An intervention group (Experimental): An intervention group: will include 41 patients who will receive the oral care bundle.
  Interventions: Procedure: oral care bundle implementation
- A control group (No Intervention): A control group: will include 41 patients who will receive the traditional oral care.

INTERVENTIONS:
Procedure: oral care bundle implementation — oral care bundle encompasses oral assessment, tooth brushing, oral / lip moisturization, and suctioning oropharyngeal secretions above the cuff.
  Arms: An intervention group

SUMMARY:
Oral care is a fundamental aspect of nursing that impact the health and comfort of patients over both the short and long term. Caring for very sick patients in a busy stressful environment may result in oral care having a lower priority for nurses than other aspects of care (Sarangi, Simon, & Sarangi, 2021). Negligence of these interventions can cause long-term oral problems and nosocomial diseases most notably VAP (Abd Alraheem, 2020).

A study conducted by Ayşe et al. (2019) reported that the application of regular oral care for the MV patients as a part of care protocols decreased bacterial colonization and had a protective and improving effect on oral health. A recent study conducted by Rizk, Saad-eldeen and Helmy (2020) concluded that VAP is a serious ICU acquired infection with significant impact and required effective preventive action. A systematic review conducted by Kharel, Bist and Mishra (2021) concluded that VAP is a critical issue in ICU with a high-cost burden and various interventional educational programs like staff training and hygiene awareness can reduce the future risk of VAP.

A recent study conducted by Abd Alraheem (2020) illustrated that 53.3% of the MV patients had average oral alteration. Asystematic review conducted by Kharel et al. (2021) to assess VAP among ICU patients in WHO South east Asian region illustrated that the VAP incidence rate ranged from 0.2% to 11.6% differing greatly between countries. The highest VAP prevalence rate was reported from the medical ICU, India, where as the lowest was from the palliative care ICU, South Korea.

In Egypt, analysis of VAP was done in some Egyptian University Hospitals by Fathy, Abdelhafeez, EL-Gilany and Abd Elhafez, (2013) who reported that the incidence of VAP ranged from 16% to 75%, the lowest ratio was in Alexandria University 16% and the highest one in Ain Shams University 75%. The incidence in Mansoura University Hospitals (MUH) was 22.6%. Another recent study conducted by Elkolaly, Bahr, El-Shafey, Basuoni, and Elber (2019) reported that the incidence of VAP in Tanta University Hospitals is still high (38.4%).

Many studies investigated the effect of oral care with chlorhexidine on the incidence of VAP and oral health in MV patients (Abd Alraheem, 2020; Collins et al., 2020; Heck, 2012; Moustafa, Tantawey, El-Soussi and Ramadan, 2016; Plantinga et al., 2016). However, the recent reappraisal of the evidence suggests that chlorhexidine does not reduce VAP, causes excess mortality in non-cardiac surgery patients (Dale et al., 2019) and unexpected high incidence of oral mucosal lesions (Plantinga et al., 2016).

Moreover, from my empirical experience, chlorhexidine is not available in all Egyptian hospitals because of its economic burden. A study conducted by Moustafa et al. (2016) recommended regular updates about evidence-based guidelines for oral care and its effect on VAP prevention and oral health. The debate of the literature about oral care inspired us to investigate this area.

DETAILED DESCRIPTION:
Critically ill patients admitted to the intensive care units (ICUs) frequently require ventilatory support as a life-saving therapy (Modrykamien, 2019). Mechanical ventilation (MV) is required for those patients as their ability to breathe is impaired secondary to trauma, recent surgery, or a medical condition (Zhao et al., 2020). Ventilation is provided via tracheal intubation which can be an entry point and place of bacteria colonization and causes many complications such as ventilator-associated pneumonia (VAP) and oral infections (Anggraeni, Hayati, &Nur'aeni, 2020).

Ventilator-associated pneumonia is a serious healthcare-associated infection (Hellyer, Ewan, Wilson, & Simpson, 2016). It is defined as a lung infection that develops in a person who is on a ventilator for more than 48 hours (Centers for Disease Control and Prevention, 2010). It can cause increased mortality and morbidity, and consequently, increased health-related costs (Wu, Wu, Zhang, & Zhong, 2019). A study conducted by Othman and Abdelazim (2017) revealed that ventilation time and ICU length of stay (LOS) were significantly longer in patients with VAP than in those without VAP.

Recent evidence has challenged widespread practices to prevent VAP such as elevating the head of the bed, implementing daily sedation holds, and effective oral hygiene. Such interventions are often used within a bundle of care (Hellyer et al., 2016). According to Institute for Health Care Improvement (IHI, 2021), the bundle of care is a structured way of improving the processes of care and patient outcomes which includes a small, straightforward set of three to five evidence-based practices that should be performed collectively and reliably.

According to the World Health Organization (WHO, 2021), oral health is a state of being free from mouth and facial pain and oral diseases that limit an individual's capacity in biting, chewing, smiling, speaking, and psychosocial well-being. A prospective cohort study conducted by Shiraishi et al. (2018) investigated the association between impaired oral health status on admission and poor clinical outcomes in post-acute inpatients. They revealed that patients with oral health problems had a significantly longer LOS and higher mortality rate than patients without oral health problems.

Oral care is a preventive and cost-effective practice for patients, particularly those who are mechanically ventilated. It helps the patient to maintain the cleanliness of his mouth and to encourage the flow of saliva that maintains a healthy oropharyngeal mucosa (Emery, & Guido-Sanz, 2019). The implementation of effective oral care can reduce the incidence of VAP (Wei, & Yang, 2019) and control the accumulation of oral pathogens (Rumagihwa, & Bhengu, 2019).

Critically ill patients are dependent on hospital staff to meet their needs for nutrition and hygiene, including oral hygiene (Zhao et al., 2020). Hence, critical care nurses (CCNs) as caregivers have an important role in providing oral care to maintain oral health and prevent infection (Anggraeni et al., 2020). The skills to provide effective oral care are available, but CCNs seem to have difficulties in translating these components into practice (Andersson, Wilde-Larsson,&Persenius, 2018).

In Egypt, a recent study conducted by Abd Alraheem (2020) to assess the effect of oral hygiene for patients on mechanical ventilation in ICU reported that about three-quarters of CCNs had an incompetent level of practice regarding oral hygiene. Meanwhile, it was found that about half of the MV patients had average oral alteration, and there was a significant relationship between oral alteration and the frequency of oral care. Another recent study conducted by da Silva Junior et al. (2020) concluded that although the nursing staff perceives oral hygiene as a part of essential patient care; still, oral hygiene practices have been neglected.

The standardized and consistent oral care practices have been successful in preventing hospital-acquired infections, most notably VAP (DeVaul, 2020). CCNs should implement evidence-based interventions that can decrease the LOS of ICU, hospital costs and protect the patients from VAP infection (Hellyer et al., 2016). A study conducted by Heck (2012) about decreasing VAP in the ICU: a sustainable comprehensive quality improvement program and revealed that the oral care bundle has proven to be a sustainable method for VAP prevention as the VAP rate per 1,000 ventilator days dropped significantly from 10.5 to 0 (P= 0.16). According to Dale et al. (2019), it encompasses oral assessment, tooth brushing, oral / lip moisturization, and suctioning oropharyngeal secretions above the cuff.

All critically ill patients should be assessed using a standardized oral care assessment tool to ensure consistency between the caring staff and reduce the incidence of nosocomial pneumonia (Collins et al., 2020). Tooth brushing is critical to maintain good oral health (Raison, Corcoran, Burnside, & Harris, 2020). Physical brushing of the teeth will remove plaque and bacteria which may reduce VAP and promote patient comfort (Collins et al., 2020). A study carried out by Ayşe, Karahan, and Cömert (2019) recommended using soft tooth brushes to remove dental plaques and maintain oral hygiene among the patients on mechanical ventilatory support.

A systematic review by de Camargo, da Silva, and Chambrone (2019) reported that all studies evidenced the importance of oral health measures in preventing VAP among MV patients. Another study conducted by Collins et al. (2020) presented that ICUs need to ensure that policies and practices are in place to promote effective oral care programs. In addition, health care professionals need to be provided with education and training to ensure compliance with it.

Finally, oral care for MV patients has developed from being a matter of patient comfort to be a matter of VAP and oral infection prevention. If the benefits of oral care outweigh the risks, accurate oral care procedures should be considered an essential and crucial component of critical care nursing. Hence, this study will be carried out to determine the effect of implementing an oral care bundle on CCNs' practice and MV patients' outcomes.

Significance of the study Oral care is a fundamental aspect of nursing that impacts the health and comfort of patients over both the short and long term. Caring for very sick patients in a busy stressful environment may result in oral care having a lower priority for nurses than other aspects of care (Sarangi, Simon, & Sarangi, 2021). Negligence of these interventions can cause long-term oral problems and nosocomial diseases most notably VAP (Abd Alraheem, 2020).

A study conducted by Ayşe et al. (2019) reported that the application of regular oral care for the MV patients as a part of care protocols decreased bacterial colonization and had a protective and improving effect on oral health. A recent study conducted by Rizk, Saad-eldeen, and Helmy (2020) concluded that VAP is a serious ICU acquired infection with significant impact and required effective preventive action. A systematic review conducted by Kharel, Bist, and Mishra (2021) concluded that VAP is a critical issue in ICU with a high-cost burden, and various interventional educational programs like staff training and hygiene awareness can reduce the future risk of VAP.

A recent study conducted by Abd Alraheem (2020) illustrated that 53.3% of the MV patients had average oral alteration. A systematic review conducted by Kharel et al. (2021) to assess VAP among ICU patients in the WHO Southeast Asian region illustrated that the VAP incidence rate ranged from 0.2% to 11.6% differing greatly between countries. The highest VAP prevalence rate was reported from the medical ICU, India, whereas the lowest was from the palliative care ICU, South Korea.

In Egypt, analysis of VAP was done in some Egyptian University Hospitals by Fathy, Abdelhafeez, EL-Gilany, and Abd Elhafez, (2013) who reported that the incidence of VAP ranged from 16% to 75%, the lowest ratio was in Alexandria University 16% and the highest one in Ain Shams University 75%. The incidence in Mansoura University Hospitals (MUH) was 22.6%. Another recent study conducted by Elkolaly, Bahr, El-Shafey, Basuoni, and Elber (2019) reported that the incidence of VAP in Tanta University Hospitals is still high (38.4%).

Many studies investigated the effect of oral care with chlorhexidine on the incidence of VAP and oral health in MV patients (Abd Alraheem, 2020; Collins et al., 2020; Heck, 2012; Moustafa, Tantawey, El-Soussi and Ramadan, 2016; Plantinga et al., 2016). However, the recent reappraisal of the evidence suggests that chlorhexidine does not reduce VAP, causes excess mortality in non-cardiac surgery patients (Dale et al., 2019), and unexpected high incidence of oral mucosal lesions (Plantinga et al., 2016).

Moreover, from my empirical experience, chlorhexidine is not available in all Egyptian hospitals because of its economic burden. A study conducted by Moustafa et al. (2016) recommended regular updates about evidence-based guidelines for oral care and its effect on VAP prevention and oral health. The debate of the literature about oral care inspired us to investigate this area.

Aim of the study This study aims to investigate the effect of implementing oral care bundle on CCNs' practice and MV patients' outcomes.

Research Hypotheses

To fulfill the aim of this study, the following research hypotheses are formulated:

* H1: The implementation of oral care bundle will enhance the CCNs' practice.
* H2: Mechanically ventilated patients who receive an oral care bundle will have a better outcome than those who receive routine hospital oral care.

Operational Definition

Patients' Outcomes:

In the context of this study patients' outcomes includes:

* Oral Health: normal oral health.
* Ventilator-Associated Pneumonia: low VAP rates.

Methods Design A quasi-experimental research design with a nonequivalent control group pretest-posttest type will be utilized in this study. It involves comparing two or more groups of people before and after implementing an intervention without randomization (Polit, & Beck, 2018).

Setting This study will be conducted at the Surgical Intensive Care Units (SICUs) at Mansoura Emergency Hospital. There are three SICUs, each one has 10 beds and provides care to patients with neurological problems and multiple trauma injuries. These units are well equipped with advanced technology and manpower required for patients' care. The nurse-patient ratio in these units is nearly 1:2.

Subjects

The subjects of this study include a pair of groups as follows:

1. Nurses: The study involves a convenience sample of nurses working in the previously selected ICUs who have more than 6 months of working experience, applying direct patient care, and accept to participate in the investigation.
2. Patients: This investigation will also include a convenience sample of 82 patients necessitating invasive mechanical ventilation and agree to participate in the study. These patients will be divided randomly into two groups:

   * An intervention group: will include 41 patients who will receive the oral care bundle.
   * A control group: will include 41 patients who will receive traditional oral care.

Patient sample size calculation

Based on data from the literature (Karkada, 2015), considering the level of significance = 5%, Power = 80%, Type of test = two-sided, Formula of calculating sample size is:

n = [2(Zα/2 + Zβ)2 × p (1-p)]/(p1 - p2)2

* n = sample size required in each group,
* p = pooled proportion (proportion of event in group 1 + proportion of event in group 2)/2
* p1-p2 = difference in proportion of events in two groups
* Zα/2: This depends on level of significance, for 5% this is 1.96
* Zβ: This depends on power, for 80% this is 0.84
* n = [2(1.96 + 0.84)2 × 0.55 (1-0.55)]/(0.31)2=40.4
* Based on the above formula, the sample size required per group is 41.

Inclusion criteria

* Adult patient > 18 years old.
* Orally intubated mechanically ventilated patients for at least 48 hours.

Exclusion criteria

Patients will be excluded from the study if they have:

* A clinical diagnosis of pneumonia at the time of admission and/or a modified Clinical Pulmonary Infection Score of 6 or greater.
* Contraindication to oral care intervention such as severe oral trauma, oral ulcerations, facial fractures, or unstable cervical fractures.

Tools Two tools will be utilized to collect data pertinent to this study. Tool I: Nurses' Practice of Oral Care Bundle Observation Checklist

It will be used pre and post-implementation of the oral care bundle. It includes two parts:

Part I: Nurses' demographic characteristics This part will be developed by the primary investigator (PI). It will include the demographic characteristics of the participant nurses' as age, gender, educational level, shift time, years of work experience in ICU, and attending previous in-service training courses or programs about oral care bundle.

Part II: Oral care bundle observation checklist This part will be developed by PI after revising related literature (Barnason et al., 1998; Collins et al., 2020; Dale et al., 2019; da Silva Junior et al., 2020; DeToye, 2019; Odgaard, & Kothari, 2019; Rumagihwa,& Bhengu, 2019). It will be used to assess nurses' practice regarding the implementation of the oral care bundle which encompasses four interventions: oral assessment, tooth brushing, oral/lip moisturization, and suctioning oropharyngeal secretions above the cuff.

Scoring system: The intervention that is done correctly will be scored with 1 point while the item that is done incorrectly or not done will be scored with zero point. The total scoring will be classified into two categories as follows:

* Satisfactory level of practice: > 80 %
* Unsatisfactory level of practice: < 80%

Tool II: Mechanically Ventilated Patients' Outcomes Evaluation Sheet

This tool will include three parts:

Part I: Patients' characteristics and health-relevant data This part will be developed by PI. It aims to assess patients' characteristics and health-relevant data. It will include patients' age, gender, smoking history, diagnosis, past medical history, total LOS in ICU, and intubation duration.

Part II: VAP diagnostic criteria sheet This part will include the modified Clinical Pulmonary Infection Score (CPIS) which will be adopted from Singh, Rogers, Atwood, Wagener, and Yu (2000) for the clinical diagnosis of VAP. This is a standard scale based on five clinical items, each scored 0-2 points including body temperature, tracheal secretion, blood leukocytes, oxygenation (calculated as PaO2 divided FiO2) and chest radiography infiltrates.

Part III: Oral assessment scale This part will be adopted from Barnason et al. (1998) to assess the oral health status of intubated patients. The oral assessment scale is composed of 6 items including the lips, tongue, saliva, mucous membrane, gums, and teeth. According to Moustafa et al. (2016), content validity for this scale has been established and it has a high reported interrater reliability (r=0.91). Each item has 3 subitems and the total scores ranged from 6 to 18.

Pilot Study A pilot study will be carried out on 10% of the total sample (patients and nurses), who will be excluded from study subjects. It will be conducted to test the feasibility and clarity of the tools. Necessary modifications will be done accordingly.

Data Collection This study will be conducted in three phases; preparation, implementation, and evaluation.

1. Preparation phase

   * Ethical approval will be obtained from the Research Ethics Committee (REC) of the Faculty of Nursing - Mansoura University.
   * Permission to conduct the study will be obtained from the responsible authorities of the study setting after explaining the aim and procedure of the study.
   * Content validity of the tool I will be reviewed by a panel of five experts in the study field and the suggestions of the jury members will be considered.
   * The reliability of tool I will be assessed using Cronbach's Alpha Test.
2. Implementation phase The PI will assess and evaluate nurses' practice and patients' outcomes in two phases as follow: pre-intervention and immediately post-intervention.

   * For nurses:

     * The PI will introduce herself to the nurses, explain the aim and nature of the study and invite them to participate in the study.
     * Nurses' demographic characteristics will be collected by using part I of tool I.
     * Critical care nurses' practice of the oral care bundle will be observed by using part II of tool I.
   * For patients:

     * An initial assessment will be carried out for all MV patients in selected ICUs on admission to confirm that they are free from exclusion criteria.
     * Patients' characteristics and health-relevant data will be collected by the PI on the first day of admission using part I of tool II.
     * Assessment of the occurrence of VAP will be done for both groups on the first, third, and sixth days of the patient's admission to the ICU by using part II of tool II.
     * An oral assessment scale will be carried out for both groups on the first, third, and sixth days of patient admission by using part III of tool II.
     * The PI will use a non-participant observation approach in collecting the data to maintain distance, no interaction, and conceal her role to avoid bias.
   * Designed booklet

     * Based on reviewing the recent related literature (Dale et al., 2019; da Silva Junior et al., 2020; DeToye, 2019; Rumagihwa, & Bhengu, 2019), the researcher will design a booklet to review the core components of the oral care bundle.
     * The initial draft of the constructed booklet will be disseminated to expertise in the field to assess its content validity. Any specific comments and recommended modifications will be considered in the formulation of the final booklet draft.
     * The booklet will be translated into Arabic after performing the back-translation technique.
     * The nurses will be educated about the content of the designed booklet in the form of lectures within 4 weeks or more according to nurses' needs (2 sessions/ week). Every session will last for about 30 minutes.
     * Each trained nurse will receive a hard copy of the designed booklet to ensure the continuity of patient care.
3. Evaluation phase

This phase aims to:

* Evaluate the effect of implementing an oral care bundle on CCNs' practice using tool I and MV patients' outcomes using tool II.
* Compare the obtained patient and nurses data pre and post-implementation of oral care bundle practices.

Data Analysis Data will be analyzed using the Statistical Package of Social Sciences (SPSS) version 21.0. It will be computerized and analyzed using appropriate descriptive and inferential statistical tests. Statistical analysis will be done according to the most current reliable and valid statistical methods.

Ethical Considerations Ethical approval will be obtained from the REC of the Faculty of Nursing - Mansoura University. Permission to conduct the study will be obtained from the hospital's administrative authority after providing a complete explanation of the aim and nature of the study. Written informed consent will be obtained from the study samples (patients' next of kin & nurses) after providing them with details about the nature of the study including the aim, procedure, benefits, and risks. They will be informed that participation in the study is voluntary and that they have the right to withdraw at any time without any responsibility. They will be also assured that their data will be coded, and their personal information will be kept confidential. There will be no link between their personal information and published data. The participant nurses will be assured that the observed practice is not a part of their annual appraisal.

ELIGIBILITY:
Inclusion criteria

* Adult patient > 18 years old.
* Orally intubated mechanically ventilated patients for at least 48 hours.

Exclusion criteria

Patients will be excluded from the study if they have:

* A clinical diagnosis of pneumonia at the time of admission and/or a modified Clinical Pulmonary Infection Score of 6 or greater.
* Contraindication to oral care intervention such as severe oral trauma, oral ulcerations, facial fractures, or unstable cervical fractures.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
oral health | one week
  The oral assessment scale will be used to assess the oral health. It is composed of 6 items including the lips, tongue, saliva, mucous membrane, gums, and teeth.

SECONDARY OUTCOMES:
Ventilator associated pneumonia | one week
  the modified Clinical Pulmonary Infection Score (CPIS) is a standard scale based on five clinical items, each scored 0-2 points including body temperature, tracheal secretion, blood leukocytes, oxygenation (calculated as PaO2 divided FiO2) and chest radiography infiltrates.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Emergency Hospital, Al Mansurah, Dakahlia Governorate, Egypt